CLINICAL TRIAL: NCT00685152
Title: High Frequency Repetitive Transcranial Magnetic Stimulation (rTMS) in the Treatment of Post-traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Roumen Milev, Professor of Psychiatry and Psychology, Head, Department of Psychiatry Queen's University, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: psiy-267-07
Record Dates: First submitted 2008-05-08; First posted 2008-05-28 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Post-Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active rTMS (Experimental): Repetitive Transcranial Magnetic Stimulation
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS) (MagPro, Medtronic)
- 2 (Sham Comparator): Device: Sham (placebo)
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS) (MagPro, Medtronic)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) (MagPro, Medtronic) — 6 weeks of either Active or Sham Repetitive Transcranial Magnetic Stimulation (rTMS). Active treatment comprises of stimulation with rTMS frequency 20Hz, intensity 110% of Motor Threshold, 20 trains, 9 seconds per train, 51 seconds of intertrain interval that is applied over the Right Dorsolateral Prefrontal Cortex by a figure eight shaped coil. Treatment will be given 5 times a week for 4 weeks, 3 times a week during Week 5 and 2 times a week during Week 6. Sham treatment will mimic active treatment; The rTMS machine used is MagPro and the company name is Medtronic.
  Other Names: rTMS machine (MagPro, Medtronic).

SUMMARY:
This is a double-blind, randomized, placebo-controlled study evaluating the efficacy and safety of high-frequency (20Hz) rTMS applied to the right dorsolateral prefrontal cortex for 6 weeks. The primary objective is to evaluate the change in PTSD symptoms before and after six weeks of high-frequency rTMS treatment as measured by the Clinician Administered PTSD Scale (CAPS) in both active and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Signed Patient Information and Consent.
* Patients with primary Post-Traumatic Stress Disorder (as diagnosed by MINI) and DSM IV TR.
* Patients with CAPS score of at least 40.
* Males or females between 18-65 years of age.
* Patients not taking PTSD pharmacotherapy for at least last 2 weeks prior to commencing in the study or if they are taking PTSD pharmacotherapy it must be stable for at least 6 weeks prior to the start and not be changed during the 6 weeks of the study treatment phase.
* Individual or group supportive psychotherapy may continue during the study but will not be allowed to start new psychotherapy during the 6 weeks of the study treatment phase.

Exclusion Criteria:

* Current primary Axis I disorder including Schizophrenia, Bipolar Disorder type I, Major Depressive Disorder.
* Other primary Axis I disorders which, in the opinion of the investigator, may affect the outcome of this study.
* Patients with HDRS score ≥ 18.
* A metallic implant in cranium (except the mouth).
* Patients with severe or unstable medical conditions, which in the opinion of the investigator would interfere with their progress or safety.
* ECT treatment within the last three months.
* Patients with a history of epilepsy.
* Patients with neurological disorder leading to increased intracranial pressure.
* Patients with severe cardiac disorder or intracardiac lines and pacemakers.
* Patients with current suicide risk ≥ 6 points by MINI.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS) in both active and sham groups | pre, week 2,4,6,8 & 12

SECONDARY OUTCOMES:
Treatment Outcome PTSD scale (TOP-8) | Pre, week 2,4,6,8 & 12
Hamilton Anxiety Scale | Pre, week 2,4,6,8 & 12
Hamilton Depression Rating Scale | Pre, week 2,4,6,8 & 12
Clinical Global Impression Scale (both severity and improvement) | Pre, week 2,4,6,8 & 12
Social Functioning-36 Quality of Life Scale version(1) | Pre, week 2,4,6,8 & 12
Pittsburgh Sleep Quality Index | Pre, week 2,4,6,8 & 12
PTSD Checklist-civilian (PCL-C) | Pre, week 2,4,6,8 & 12

CONTACTS AND LOCATIONS:
Overall Officials: Roumen Milev, MD, Principal Investigator — Queen's University
Locations (2):
- Dr. Dancho Dilkov, Sofia, Bulgaria
- Providence Care Mental Health Services, Kingston, Ontario, Canada